CLINICAL TRIAL: NCT01259336
Title: A RANDOMIZED CONTROLLED STUDY OF ITRACONAZOLE IN CHRONIC CAVITARY PULMONARY ASPERGILLOSIS
Brief Title: Efficacy Of Itraconazole In Chronic Cavitary Pulmonary Aspergillosis
Acronym: ITRACONASP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vishwanath gella, vgella, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Itracon asp
Record Dates: First submitted 2010-12-06; First posted 2010-12-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Cavitary Pulmonary Aspergillosis
Keywords: Itraconazole; chronic cavitary pulmonary aspergillosis; Aspergillosis; fungal ball; mycetoma; efficacy; safety
MeSH Terms: conditions — Aspergillosis; Mycetoma | interventions — Itraconazole; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itraconazole (Active Comparator): Role of itraconazole in CCPA
  Interventions: Drug: Itraconazole; Drug: treatment in cavitary pulmonary aspergillosis
- treatment in cavitary pulmonary aspergillosis (Experimental): Patients in this arm are given conservative management with antitussives, brochial artery embolisation.
  Interventions: Drug: treatment in cavitary pulmonary aspergillosis

INTERVENTIONS:
Drug: Itraconazole — Tablet 200 mg twice daily for 6 months
  Other Names: Study group
  Arms: Itraconazole
Drug: treatment in cavitary pulmonary aspergillosis — Anti-tussive, blood transfusion, surgical resection and bronchial artery embolisation(BAE)

SUMMARY:
The purpose of this study is to determine whether there itraconazole is effective in the treatment of chronic cavitary pulmonary aspergillosis

DETAILED DESCRIPTION:
The role of itraconazole is still not clear in the treatment of chronic cavitary pulmonary aspergillosis(CCPA). Some studies have shown a beneficial role of itraconazole in reducing hemoptysis. So the present study is aimed at analyzing the role of itraconazole in CCPA.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Clinical symptoms: -presence of chronic pulmonary/systemic symptoms lasting ≥ six weeks.
   2. Radiological findings:

      * Evidence of slowly progressive pulmonary lesions over weeks-months including cavities with surrounding inflammation.
      * presence of intracavitary mass with a surrounding crescent of air,and presence of pleural thickening in peripheral lesions.
   3. Microbiological/Immunological findings: Positive results in the aspergillus precipitin test, demonstration of aspergillus hyphae in sputum or BAL fluid or cultures of BAL/sputum growing aspergillus species.
2. The diagnosis of CCPA will be made if

   1. Patient satisfies at least 1, 2a or 2b and/ or any of the 3rd criteria.
   2. FNAC from the cavity wall will be considered in atypical cases
3. Exclusion Criteria:

   1. Invasive aspergillosis
   2. Allergic broncho-pulmonary aspergillosis (ABPA)
   3. Active tuberculosis or malignancy
   4. Pregnant females

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
clinical improvement in cough and hemoptysis | 6 months
  Clinical response- assessed by a decrease in frequency & intensity of hemoptysis & cough. Significant clinical response will be considered if there is no recurrence of episodes of moderate-massive hemoptysis. Number of interventions required to control hemoptysis will also be taken as a measure of clinical response

SECONDARY OUTCOMES:
Radiological response of CCPA to itraconazole | 6 months
  1. Complete response- It is defined as complete disappearance of the aspergilloma.
  2. Partial response- It is defined as 30% decrease in the sum of the longest diameters of all the lesions.
  3. Progressive disease- It is defined as appearance of any new lesions or >20% increase in the sum of the longest diameters of all measurable lesions.
  4. Stable disease- Shrinkage or growth of CCPA that does not meet any of these criteria

CONTACTS AND LOCATIONS:
Overall Officials: Vishwananath gella, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Punjab, India

REFERENCES:
- [Background] Stevens DA, Kan VL, Judson MA, Morrison VA, Dummer S, Denning DW, Bennett JE, Walsh TJ, Patterson TF, Pankey GA. Practice guidelines for diseases caused by Aspergillus. Infectious Diseases Society of America. Clin Infect Dis. 2000 Apr;30(4):696-709. doi: 10.1086/313756. Epub 2000 Apr 20. PMID 10770732
- [Derived] Agarwal R, Vishwanath G, Aggarwal AN, Garg M, Gupta D, Chakrabarti A. Itraconazole in chronic cavitary pulmonary aspergillosis: a randomised controlled trial and systematic review of literature. Mycoses. 2013 Sep;56(5):559-70. doi: 10.1111/myc.12075. Epub 2013 Mar 18. PMID 23496375